CLINICAL TRIAL: NCT05615103
Title: The Efficiency of 18F-FDG PET-CT for Predicting Advanced Oesophageal Squamous Cell Carcinoma Patients' Tumor Response to Immunochemotherapy in the Neoadjuvant Setting
Brief Title: The PET-CT Predicting Response to Immunochemotherapy in Esophageal Cancer
Acronym: POSITRON
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Guangdong Provincial People's Hospital (Other)
Collaborators: First Affiliated Hospital of Shantou University Medical College (Other); Shenzhen People's Hospital (Other); The Affiliated Cancer Hospital of Guangzhou Medical University (Unknown)
Responsible Party: Sponsor
Other Study IDs: POSITRON
Record Dates: First submitted 2022-11-07; First posted 2022-11-14 (Actual); Last update posted 2022-11-29 (Actual); Status verified 2022-11

CONDITIONS: Esophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Treatment with immune checkpoint inhibitors such as programmed death receptor 1 (PD-1 inhibitors) for advanced and metastatic esophageal squamous cell carcinoma (ESCC) significantly improves patients' overall survival compared to chemotherapy alone. Despite this milestone breakthrough, immunochemotherapy also has known limitations. Indeed, only 45-72% of patients achieved objective responses. It is urgent to find out easily-determined and convenient biomarkers to identify patients who will benefit from such treatment modality. Due to the luminal structure of the esophagus, the exact diameter of esophageal tumor cannot be precisely measured per RECIST 1.1. Moreover, the definition of the metastatic lymph node in which the short-axis lengths should be longer than 1.5 cm hinders the risk of missing the smaller metastatic lymph node foci. Thus, it is difficult to implement morphology-based criteria for evaluating the neoadjuvant immunochemotherapy response. The current study aimed to investigate the role of iPERCIST in predicting tumor response and the short-term overall survival of patients with locally advanced ESCC after neoadjuvant immunochemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* pathologically confirmed locally advanced ESCC (cT3-4anyNM0) that was potentially resectable after neoadjuvant immunochemotherapy.
* treatment-naïve and had the adequate cardiopulmonary function

Exclusion Criteria:

* previous autoimmune disease
* unable to complete planned treatment courses and no complete follow-up PET-CT scan

Ages: 18 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible patients were selected according to the following criteria: pathologically confirmed locally advanced ESCC (cT3-4anyNM0) that was potentially resectable after neoadjuvant immunochemotherapy. All patients were treatment-naïve and had adequate cardiopulmonary function. The exclusion criteria included previous autoimmune disease; unable to complete planned treatment courses and no complete follow-up PET-CT scan.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-11-08 (Actual); Primary Completion 2023-09-08 (Estimated); Study Completion 2023-12-08 (Estimated)

PRIMARY OUTCOMES:
Pathologic complete response rate (pCR) | Three to five working days after surgery
  The rate of pathologic complete response rate after the combined treatment of chemotherapy and immunotherapy following surgery

SECONDARY OUTCOMES:
Overall survival | from the date of diagnosis to the date of death, assessed up to 100 months
  Overall survival rate
Event-free survival | from the date of treatment initiation to the date of first progression (local recurrence of tumor or distant metastasis) or death from any cause, assessed up to 100 months
  EFS
Safety as measured by number of participants with Grade 3 and 4 adverse events | Up to 12 weeks
  Number of Grade 3 and 4 adverse events as defined by CTCAE v5.0

CONTACTS AND LOCATIONS:
Locations (1):
- Guangdong Provincial People's Hospital, Guangzhou, Guangdong, China